CLINICAL TRIAL: NCT05272072
Title: Evaluation of Relationship Between Preoperative Fibrinogen/Albumin Ratio and Morbidity After Hip Fracture Operations in Oldest Old Patients: A Prospective Observational Study
Brief Title: Evaluation of Relationship Between Preoperative Fibrinogen/Albumin Ratio and Morbidity After Hip Fracture Operations
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nur Canbolat, Principal Investigator, M.D., Istanbul University
Other Study IDs: 2021/1968
Record Dates: First submitted 2022-02-11; First posted 2022-03-09 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Hip Fractures; Albumin; Fibrinogen; Scoring Systems; Preoperative Risk Prediction; Elderly
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to the aging of populations, hip fracture operations are increasing from year to year. This operations have many complications also high morbidity and the mortality. Population of this study is oldest old age patients who will have an operation because of hip fracture.

The primary outcome of this study is evaluation of relationship between preoperative fibrinogen/albumin ratio and the morbidity after hip fracture operations. The secondary outcomes of this study is evaluation of relationships between fibrinogen/albumin ratio and mortality, length of stay in ICU, length of stay in hospital, postoperative complications, blood product consumption. The study will be completed after the records of preoperative, intraoperative data and the data of the first 30 days postoperatively in this population.

DETAILED DESCRIPTION:
Due to the aging of populations, hip fracture operations are increasing from year to year. This operations have many complications also high morbidity and the mortality. Elderly people are divided into 3 groups according to their age. Elderly people whose aged over 85 years as oldest-old. Population of this study is oldest old patients who will have an operation because of hip fracture.

The research is as a single-center, prospective observational study. The primary outcome of this study is evaluation of relationship between preoperative fibrinogen/albumin ratio and the morbidity after hip fracture operations. Age-Adjusted Charlson Comorbidity Index, Nottingham Hip Fracture Score and Clinical Frailty Scale Score will be calculated at the preoperative visit for each patient before operation. Investigators planned to use these three scores to determine morbidity.

Age-Adjusted Charlson Comorbidity Index AACCI): Age-modified version of the Charlson Comorbidity Index. Charlson Comorbidity Index predicts the ten-year mortality for a patient who may have a range of comorbid conditions for example diabetes, myocardial infarction, dementia, liver disease, lymphoma. Each comorbid condition has a separate point. 71 years old and older patients have +4 points for scoring of Age-Adjusted Charlson Comorbidity Index. The sum of the scores gives the total score. The minimum score is 4 for oldest old patients. Higher scores mean a worse outcome.

Nottingham Hip Fracture Score (NHFS) is a scoring system that reliably predicts 30 day mortality for patients after hip fracture. Development and validation of a preoperative scoring system to predict 30 day mortality in patients undergoing hip fracture surgery. To calculate the NHFS, it is necessary to calculate the abbreviated mental test score of 10 points in total. The minimum score is 3 for oldest old patients. The maximum score is 10. Higher scores mean a worse outcome.

The Clinical Frailty Scale (CFS) is a judgement-based frailty tool that evaluates specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill). Higher scores mean a worse outcome.

The secondary outcomes of this study is evaluation of relationships between fibrinogen/albumin ratio and Nottingham Hip Fracture Score, Clinical Frailty Scale Score, mortality, length of stay in ICU, length of stay in hospital, blood product consumption, postoperative complications. Postoperative complications are divided into pulmonary, cardiovascular, hepatic, renal complications, bleeding, electrolyte imbalance, wound site infections, delirium and other. Postoperative pulmonary complications (PPC) encompass almost any complication affecting the respiratory system after anaesthesia and surgery. PPCs are bronchospasm, aspiration pneumonia, atelectasis, pneumonia, pleural effusion, pneumothorax, pulmonary embolism, respiratory failure, acute respiratory distress syndrome, tracheobronchitis etc. Postoperative cardiac complications are resistant hypotension- hypertension, new onset of dysrhythmias like atrial fibrillation, acute coronary syndromes, cardiac failure, cardiogenic shock. Investigators will follow up postoperative hemogram and record amount of blood transfused to investigate bleeding. Investigators will follow up serum creatinin and urea level, use Kidney Disease Improving Global Outcomes (KDIGO) criteria for acute renal failure and note necessity of hemodialysis or hemodiafiltration.

Before the study, it was determined that at least 108 patients should be collected in the power analysis performed with the help of similar literature data. After collecting the demographic and peroperative data up to postoperative 30 days of the patients, the data will be transferred to the statistical program called SPSS and statistical analysis will be made. The investigators study does not contain any modifications other than the investigators daily routine practices.

ELIGIBILITY:
Inclusion Criteria:

* ≥85 years old patients
* Primary operation
* Undergoing hip fracture surgery
* Receiving consent from patients or guardians that they accept regional anesthesia
* Not having active infection
* American Society of Anesthesiologists (ASA) 1-4
* BMI< 40 kg/m²

Exclusion Criteria:

* Refusal regional anesthesia
* Infection on regional anesthesia application area
* Infection in the central nervous system
* Coagulopathy
* Known allergy against local anesthetics
* Severe hepatic insufficiency
* Haematologic disease
* Rheumatological disease
* Autoimmune disease

Min Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 85 years of age who will undergo hip fracture surgery, whose preoperative albumin/fibrinogen ratio is checked
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Morbidity | Preoperative (before induction of anesthesia)
  Age Adjusted Charlson Comorbidity Index will be calculated for morbidity estimation. This score predicts the ten-year mortality for a patient who may have a range of comorbid conditions. The minimum score is 4 for oldest old patients. The maximum score is 34. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Nottingham Hip Fracture Score | Preoperative (before induction of anesthesia)
  Development and validation of Nottingham Hip Fracture Score to predict 30 day mortality in patients undergoing hip fracture surgery. The minimum score is 3 for oldest old patients.The maximum score is 10. Higher scores mean a worse outcome.
Clinical Frailty Scale Score | Preoperative (before induction of anesthesia)
  A judgement-based frailty tool that evaluates specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill). Higher scores mean a worse outcome.
Mortality | Up to 30 days
  Death rate of the patients
Length of stay in ICU | Up to 30 days
  Duration of stay (days) in intensive care unit because of hip fracture
Length of stay in hospital | Up to 30 days
  Duration of stay (days) in hospital because of hip fracture from admission to discharge.
Postoperative complications | Up to discharge (up to 30 days)
  Addition of a new disease or problem after hip fracture operation.
Amount of intraoperative and postoperative blood product replacement | Up to discharge (up to 30 days)
  Amount of blood product replacement in operation room and after operation up to discharge (up to 30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Emine Dizem Sunal, MD, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)